CLINICAL TRIAL: NCT06280859
Title: Hoosier Sport: Developing and Implementing a Sustainable Campus-Community Partnership in Rural Indiana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kyle A. Kercher, Assistant Professor, Indiana University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 18784
Record Dates: First submitted 2024-02-11; First posted 2024-02-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Cardiovascular Diseases; Sedentary Behavior
MeSH Terms: conditions — Cardiovascular Diseases; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Students enrolled in physical education (PE) class will be eligible to enroll in the study, and serve as the intervention group. Those not enrolled in PE that semester will be recruited as the control group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention arm will receive the Hoosier Sport intervention 2-3 times a week (twice in PE class, and once in home room). This will involve learning new sport, exercise, and nutrition knowledge, as well as developing leadership skills.
  Interventions: Behavioral: Hoosier Sport
- Control (No Intervention): Participants in the control arm will not receive the Hoosier Sport intervention.

INTERVENTIONS:
Behavioral: Hoosier Sport — Hoosier Sport is a sport-based youth development intervention. The intervention targets physical activity levels, exercise and nutrition knowledge, and leadership skills. The intervention is delivered in person twice a week (Tue/Thu) during PE class. Each class lasts 45-minutes, and covers sport skills, and then a brief lecture and activity on exercise/nutrition/leadership skills. Additionally, once a week Hoosier Sport is delivered virtually (via Zoom) during home room for 20-minutes. This involves activities to allow the students to be active during the school-day.
  Arms: Intervention

SUMMARY:
The clinical trial aims to develop and pilot test a multilevel physical activity (PA) intervention called the Hoosier Sport program. The study follows a participatory co-design protocol involving youth, parents, and community leaders to provide direct input into the intervention's design. The ultimate goal is to contribute to health equity in the community by promoting sustainable physical activity. Hoosier Sport involves delivering enhanced physical education classes, teaching about nutrition and exercise, as well as developing leadership skills in middle school rural students.The intervention will last for 8-weeks with PE classes occur twice a week. Additionally, Hoosier Sport will create more opportunities for students to be active at school (e.g., in home room) through providing virtual classes and other activities.

ELIGIBILITY:
Inclusion Criteria:

* Has PE class the semester during Hoosier Sport-
* Parent provides informed consent

Exclusion Criteria:

* Answer yes to any question on the Physical Activity Readiness for Everybody (PARQ+)

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Feasibility of Intervention Measure (FIM) | Measured at week 0 and week 9
  How feasible the intervention was from the perspective of the participants. This is measured through questionnaire.
Acceptability of Intervention Measure (IAM) | Measured at week 0 and week 9
  How acceptable the intervention is to the participants. This is measured through questionnaire.
Intervention Appropriateness Measure (AIM) | Measured at week 0 and week 9
  How appropriate the intervention is to the participants. This is measured through questionnaire.

SECONDARY OUTCOMES:
Daily Steps of Participants | Week 1 (for 7 days), and week 9 (for 7 days)
  Accelerometers (Axivity - AX3 model) will be used to track daily steps
Daily Moderate to Vigorous Physical Activity of Participants | Week 1 (for 7 days), and week 9 (for 7 days)
  Accelerometers (Axivity - AX3 model) will be used to track daily MVPA
Heart Rate of Participants | HR will be taken at week 0 and week 9 before and following the 6-minute walk test.
  heart rate measured via a blood pressure monitor
Blood Pressure of Participants | BP will be taken at week 0 and week 9 before and following the 6-minute walk test.
  Blood pressure measured via a blood pressure monitor
Basic Psychological Needs of Participants in Intervention Environment | Assessed at week 0 and week 9
  Basic Psychological Needs and Satisfaction and Frustration scale (BPNSF). This entails feelings/perceptions of autonomy, relatedness, competence, enjoyment, satisfaction, and frustration in the study setting.
Physical Literacy of Participants | Assessed at week 0 and week 9
  the Canadian Assessment of Physical Literacy second addition (CAPL-2) will be used. A higher score on the CAPL-2 indicates higher physical literacy.
Cardiovascular Fitness Levels of Participants | Assessed at week 0 and week 9
  the 6-minute walk test will be used to assess changes in fitness. Greater distance walked in the 6 minute time frame is related to greater levels of cardiovascular fitness.
Muscular Endurance Levels of Participants | Assessed at week 0 and week 9
  The plank test will be used to assess changes in fitness. The longer the plank is held, the greater the muscular endurance of the participant.
Self-Reported Weekly Moderate to Vigorous Physical Activity of Participants | Assessed at week 0 and week 9
  The Canadian Assessment of Physical Literacy Second Edition (CAPL-2) will be used to assess self-reported weekly MVPA.
Nutrition Knowledge of Participants | Assessed at week 0 and week 9
  A survey will assess basic knowledge of nutrition. We will use knowledge of SNAP-Ed, the United State Department of Agriculture's recommended curriculum. There will be three questions, with a high score reflecting greater nutrition knowledge.
Policy, Systems, and Environmental Factors Influencing Participant Physical Activity and Nutrition Behavior. | Assessed at week 0 and week 9
  a survey will collect data on Policy, Systems and Environmental (PSE) changes using a 5 questions guided by the SNAP-Ed curriculum. Higher scores will indicate better PSE support for physical activity and healthy nutrition opportunities for the participants in their school environment.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
All individual participant data will be masked and only the PI will have access to the data.